CLINICAL TRIAL: NCT07375251
Title: TELEMACO-S: a Telemonitoring Project in Cardiology and Technology Transfer Using Telemedicine
Brief Title: TELEMACO-S: a Telemonitoring Project in Cardiology and Technology Transfer
Acronym: TELEMACO-S
Status: Enrolling by invitation | Type: Observational
Sponsor: Valentina Micheluzzi (Other)
Responsible Party: Sponsor-Investigator, Valentina Micheluzzi, MSN, RN, Azienda Ospedaliero Universitaria di Sassari
Organization: Azienda Ospedaliero Universitaria di Sassari (Other)
Other Study IDs: AO SASSARI
Record Dates: First submitted 2025-12-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure Patients
Keywords: Heart Failure; acute decompensated heart failure; wearable devices; telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with heart failure: Patients with stable heart failure

SUMMARY:
The primary objective of this research project is to prevent heart failure decompensation through a wearable-based telemonitoring system (smartwatches), with a focus on the development and validation of a multiparametric predictive score.

ELIGIBILITY:
Inclusion Criteria Age ≥ 18 years Diagnosis of stable heart failure Cognitively able to participate in the study No significant hearing impairment No significant visual impairment Sufficient ability to read and write in Italian Ownership of a smartphone with internet access

Exclusion Criteria Not fully compensated heart failure Lack of a smartphone with internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed in the heart failure outpatient clinic or previously hospitalized in hospital wards (e.g., cardiology, cardiac surgery, or internal medicine).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of hospitalizations for acute heart failure decompensation | From the start of the study (14 July 2025) until the end of follow-up (31 March 2026), assessed up to approximately 8.5 months (up to 37 weeks)
  Hospitalizations for acute heart failure decompensation assessed during the study period. Changes over time in the number of hospitalizations will be evaluated; a multiparametric score will be used to support clinical assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Sassari, Sassari, SS, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Indraratna P, Biswas U, Yu J, Schreier G, Ooi SY, Lovell NH, Redmond SJ. Trials and Tribulations: mHealth Clinical Trials in the COVID-19 Pandemic. Yearb Med Inform. 2021 Aug;30(1):272-279. doi: 10.1055/s-0041-1726487. Epub 2021 Apr 21. PMID 33882601
- [Background] Docherty KF, Buendia Lopez R, Folkvaljon F, Boer RA, Chen J, Hammarstedt A, Kitzman DW, Kosiborod MN, Langkilde AM, Reicher B, Senni M, Wilderang U, Verma S, Cowie MR, Solomon SD, McMurray JJV. Wearable Accelerometer-Derived Measures of Physical Activity in Heart Failure: Insights From the DETERMINE trials. J Card Fail. 2025 Apr;31(4):689-703. doi: 10.1016/j.cardfail.2024.10.439. Epub 2024 Nov 26. PMID 39603408
- [Background] Wettstein R, Sedaghat-Hamedani F, Heinze O, Amr A, Reich C, Betz T, Kayvanpour E, Merzweiler A, Busch C, Mohr I, Friedmann-Bette B, Frey N, Dugas M, Meder B. A Remote Patient Monitoring System With Feedback Mechanisms Using a Smartwatch: Concept, Implementation, and Evaluation Based on the activeDCM Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Nov 22;12:e58441. doi: 10.2196/58441. PMID 39365164
- [Background] Kitsiou S, Gerber BS, Buchholz SW, Kansal MM, Sun J, Pressler SJ. Patient-Centered mHealth Intervention to Improve Self-Care in Patients With Chronic Heart Failure: Phase 1 Randomized Controlled Trial. J Med Internet Res. 2025 Jan 15;27:e55586. doi: 10.2196/55586. PMID 39813671
- [Background] Golbus JR, Gosch K, Birmingham MC, Butler J, Lingvay I, Lanfear DE, Abbate A, Kosiborod ML, Damaraju CV, Januzzi JL Jr, Spertus J, Nallamothu BK. Association Between Wearable Device Measured Activity and Patient-Reported Outcomes for Heart Failure. JACC Heart Fail. 2023 Nov;11(11):1521-1530. doi: 10.1016/j.jchf.2023.05.033. Epub 2023 Jul 26. PMID 37498273
- [Background] Khandwalla RM, Birkeland K, Heywood JT, Steinhubl S, McCague K, Fombu E, Grant D, Riebman JB, Owens RL. Activity Sensors to Evaluate the Effect of Sacubitril/Valsartan on Quality-of-Life in Heart Failure: rational and design of the AWAKE-HF study. ESC Heart Fail. 2019 Dec;6(6):1313-1321. doi: 10.1002/ehf2.12514. Epub 2019 Oct 22. PMID 31638338
- [Background] Boehmer JP, Cremer S, Abo-Auda WS, Stokes DR, Hadi A, McCann PJ, Burch AE, Bonderman D. Impact of a Novel Wearable Sensor on Heart Failure Rehospitalization: An Open-Label Concurrent-Control Clinical Trial. JACC Heart Fail. 2024 Dec;12(12):2011-2022. doi: 10.1016/j.jchf.2024.07.022. Epub 2024 Oct 9. PMID 39387771